CLINICAL TRIAL: NCT01302483
Title: A Phase II, Single-Center, Randomized, Double-Blind, Active-Treatment-Controlled, Parallel-Group Study of the Efficacy of Kovacaine Nasal Spray for Anesthetizing Maxillary Teeth in Healthy Dental Patients
Brief Title: Safety and Effectiveness of Kovacaine Nasal Spray for Dental Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Ground Zero Pharmaceuticals (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SR 2-01
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Dental Anesthesia Efficacy
MeSH Terms: interventions — Tetracaine; Oxymetazoline; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Kovacaine Nasal Spray (Experimental): 3% tetracaine HCL with 0.05% oxymetazoline HCL - Delivered via 3 sprays (100 uL) in each nostril
  Interventions: Drug: 3% tetracaine HCL with 0.05% oxymetazoline HCL
- Lidocaine Injection (Active Comparator): .5 to 1 catridge of 2% lidocaine HCL with 1:100,000 epinephrine
  Interventions: Drug: Lidocaine Injection

INTERVENTIONS:
Drug: 3% tetracaine HCL with 0.05% oxymetazoline HCL — 1 sham injection along with 3 sprays of Kovacaine Nasal Spray in each nostril; a 4-minute interval between every set of sprays. The total dose of 3% tetracaine HCL with 0.05% oxymetazoline HCL was 18 mg/0.3 mg.
  Arms: Kovacaine Nasal Spray
Drug: Lidocaine Injection — Each subject received both an injection along with 3 sprays of isotonic saline sham in each nostril; a 4-minute interval between every set of sprays.
  Arms: Lidocaine Injection

SUMMARY:
The purpose of this study was to determine the safety and efficacy of Kovacaine Mist (3% tetracaine HCl with 0.05% oxymetazoline HCl) for anesthesia of the maxillary teeth for dental procedures.

DETAILED DESCRIPTION:
The primary objective of this single-center, randomized, double-blind, active-controlled, parallel-group study was to determine if Kovacaine Mist provided anesthesia of the maxillary teeth sufficient for the performance of dental procedures. Secondary objectives included a determination of whether Kovacaine Mist provided anesthesia of the soft tissue and to evaluate the safety and tolerability of Kovacaine Mist and sham injection as compared to sham nasal spray and 2% lidocaine hydrochloride with 1:100,000 epinephrine submucosal injection and as determined by changes in vital signs and reports of side effects and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age
* Sufficiently healthy as determined by the investigator to receive the test and control medications and undergo the scheduled dental procedure
* Required an operative restorative procedure on a single maxillary tooth, other than a maxillary second or third molar, with treatment time not expected to exceed 60 minutes
* Could breathe through both nostrils
* Had normal lip, nose, eyelid, and cheek sensations
* Could understand and sign the informed consent document
* Could communicate with the investigator
* Could understand and comply with the requirements of the protocol

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, cardiovascular, psychiatric, musculoskeletal, neurologic, genitourinary, infective, inflammatory, immunological, dermatological, or connective tissue disease or disorder or a clinically relevant history or presence of angle-closure glaucoma
* Clinically relevant sinus/nasal surgical history
* Baseline Visual Analog Scale value of > 36 (or greater than weak) at the treatment site
* Had not had dental work requiring a local anesthetic within the last 24 hours or had taken pain medications within the last 48 hours
* Required prophylactic antibiotics for subacute bacterial endocarditis (infectious endocarditis)
* Allergic to or intolerant of tetracaine, benzocaine, other ester local anesthetics, or p-aminobenzoic acid (PABA), as found in PABA-containing sunscreens
* Allergic to or intolerant of oxymetazoline, epinephrine, or preservatives in their solutions
* Had a current condition, such as nasal congestion or sinus infection, that may have influenced responses to study medications
* History of alcoholism and/or drug abuse
* Had taken a monamine oxidase inhibitor within the past 3 weeks
* Were nursing, pregnant, suspected of being pregnant, or trying to become pregnant (females were required to take a urine pregnancy test to rule out pregnancy)
* Had used any investigational drug and/or participated in any clinical trial within 30 days of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian G Ciancio, DDS, Principal Investigator — Department of Periodontics & Endodontics, School of Dental Medicine, University at Buffalo, SUNY
Locations (1):
- University of Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Ciancio SG, Hutcheson MC, Ayoub F, Pantera EA Jr, Pantera CT, Garlapo DA, Sobieraj BD, Almubarak SA. Safety and efficacy of a novel nasal spray for maxillary dental anesthesia. J Dent Res. 2013 Jul;92(7 Suppl):43S-8S. doi: 10.1177/0022034513484334. Epub 2013 May 20. PMID 23690356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed within the month of December, 2008. Subjects were primarily recruited from University of Buffalo staff and students.
Groups:
- Kovacaine Nasal Spray: .6mL 3% tetracaine HCL with 0.05% oxymetazoline HCL
- Lidocaine Injection: 2% lidocaine HCL with 1:100,000 epinephrine
Period: Overall Study
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 15 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.8) | 40.8 (15.3) | 39.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Pulpal Anesthesia
Description: Number of participants who did not need rescue anesthesia to complete the study dental procedure, i.e. Kovacaine provided enough pulpal anesthesia to complete a dental procedure.
Time Frame: Continuous throughout dental treatment period (up to 60 minutes)
Population: Intention to treat
Measure: Number; unit: participants
Groups:
- Kovacaine Nasal Spray; Lidocaine Injection: Number of subjects able to complete the dental procedure without rescue
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Number analyzed (Participants) | 30 | 15
participants | 25 | 14

2. Secondary Outcome: Soft Tissue Anesthesia Duration
Description: Assessment of pain using a Rotadent sensor probe, applying up to 20 grams/cm^2 at the tissue site. At each time point, participants were asked if they felt pain from the sensor probe at each site location in the mouth. The four sites were:
  * Site 1: Distal to the apex of the tooth in the position of the maxillary first premolar at the deepest point in the buccal vestibule
  * Site 2: Apical to the maxillary lateral incisor at the deepest point in the labial vestibule
  * Site 3: Incisive papilla
  * Site 4: At the confluence of the alveolar process and hard palate medial to the maxillary second premolar (near the greater palatine foramen)
Time Frame: Baseline, 15, 20, 30, 40, 50, 60, 80, 100, 120 minutes
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Kovacaine Nasal Spray; Lidocaine Injection: Duration of Soft Tissue Anesthesia
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Number analyzed (Participants) | 30 | 15
Minutes
  Site 1 Duration | 21.1 (16.9) | 34.2 (21.0)
  Site 2 Duration | 16.1 (16.9) | 32.1 (4.9)
  Site 3 Duration | 31.8 (19.9) | 25.0 (18.3)
  Site 4 Duration | 31.4 (24.1) | 29.3 (27.6)

3. Secondary Outcome: Maximum Change in Pulse From Baseline
Description: Maximum change from Baseline at any time point.
Time Frame: Baseline, 15, 20, 30, 40, 50, 60, 120 minutes
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Number analyzed (Participants) | 30 | 15
beats per minute | -11.13 (9.68) | -6.60 (15.58)

4. Secondary Outcome: Maximum Change in Blood Pressure From Baseline
Description: Maximum change from Baseline at any time point.
Time Frame: Baseline, 15, 20, 30, 40 50, 60, 120 minutes
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Kovacaine Nasal Spray; Lidocaine Injection: Blood Pressure Maximum Change from Baseline
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Number analyzed (Participants) | 30 | 15
mmHG
  Systolic blood pressure | 4.50 (17.39) | 3.43 (10.62)
  Diastolic blood pressure | -2.67 (13.73) | -5.07 (8.49)

5. Secondary Outcome: Maximum Change in Pulse Oximetry From Baseline
Description: Maximum change from Baseline at any time point
Time Frame: Baseline, 15, 20, 30, 40, 50, 60, 120 minutes
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: SpO2
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Number analyzed (Participants) | 30 | 15
SpO2 | 0.17 (2.39) | -0.80 (2.76)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Kovacaine Nasal Spray | Lidocaine Injection
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 10/30 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Nasal Spray (N=30) | Lidocaine Injection (N=15)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
The VAS was misadministered such that even subjects with enough pain to require rescue reported essentially no pain on the global VAS. As this would exaggerate the efficacy of the study drug, these measures were not used to calculate its efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No